CLINICAL TRIAL: NCT01654900
Title: Mid -Term Survival and Quality of Life of Elderly Patients Undergoing Open Heart Surgery
Brief Title: Mid-term Survival and Quality of Life of Elderly Patients Undergoing Open Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Heart90-HMO-CTIL
Record Dates: First submitted 2012-07-16; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients age >75 y who underwent open hear surgeary: The cohort study consist of all patients > 75 y, undergoing open heart surgery between 2008-2011 at Hadassah medical center.
  Interventions: Other: No intervention in this study

INTERVENTIONS:
Other: No intervention in this study

SUMMARY:
The purposes of the investigators study is to examine the overall survival and quality of life in elderly patients (> 75 years) undergoing open heart surgery at Hadassah medical center between 2008-2011. All alive patients will be phone interviewed using the 36-item short form health survey. Results will be compared to similar health survey results (36-SF)obtained from a group of Israeli adults who had no open heart surgery (controlled group). The investigators hypothesize that elderly patients achieve improvement in quality of life after open heart surgery with acceptable operative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* all patients age > 75 years who discharged alive after surgery

Exclusion Criteria:

* death

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients age >75 y who underwent open heart surgery between 2008-2011 at hadassah medical center.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2012-10

PRIMARY OUTCOMES:
Quality of life | 2-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Oz Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Ein Kerem, Israel